CLINICAL TRIAL: NCT01398072
Title: A Phase III Single-blind, Randomised Placebo Controlled Trial of Long Term Therapy in Patients With Stable COPD Using Moxifloxacin, Azithromycin and Doxycycline: a Bayesian Decision Analysis, Including Other Criteria, Will be Used to Distinguish the Optimal Antibiotic Treatment
Brief Title: Development of an Optimal Antibiotic Regime for Long-term Therapy in Stable Chronic Obstructive Pulmonary Disease (COPD)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Collaborators: Royal Free Hampstead NHS Trust (Other); University of Cambridge (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Alison Evans, University College London
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 11/0078
Record Dates: First submitted 2011-07-18; First posted 2011-07-20 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2012-05

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD).
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Moxifloxacin; Azithromycin; Doxycycline

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Moxifloxacin (Active Comparator)
  Interventions: Drug: Moxifloxacin
- Azithromycin (Active Comparator)
  Interventions: Drug: Azithromycin
- Doxycycline (Active Comparator)
  Interventions: Drug: Doxycycline
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Moxifloxacin — An oral dose of 400 mg once daily for 5 consecutive days every 4 weeks.
  Arms: Moxifloxacin
Drug: Azithromycin — An oral dose of 250 mg once daily three times a week (every other day).
  Arms: Azithromycin
Drug: Doxycycline — An oral dose of 100 mg once daily.
  Arms: Doxycycline
Drug: Placebo — Oral dose of one table once daily.
  Arms: Placebo

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is the cause of considerable deaths, and exacerbations (flare up of symptoms) are a major cause of hospital admission in the UK. Bacterial infections play an important role in the development of COPD, however, there is little information available about the use of long term antibiotics in the treatment of this disease. Therefore the purpose of this study is to identify the best antibiotic regime for treating patients with COPD who have persistent bacterial infection in their lung. We will test a variety of approaches including both older and newer regimes prescribed either on a daily basis at a lower dose or in "pulsed" courses (for example, every other day or five days every month). The three antibiotics tested in this study are: moxifloxacin, azithromycin and doxycycline. This is a 13 weeks study conducted at the Royal Free Hospital, London. It is expected that approximately 200 patients will be selected for this study. The information we get from this study may help us to treat future patients with COPD better.

DETAILED DESCRIPTION:
This is a 14 week study in which 200 patients with COPD will be selected for this study from GP practices up to a 15 mile radius from the Royal Free Hospital to participate in this study. The 3 antibiotic regimes (plus a placebo group) will be used in this study are:

Moxifloxacin: an oral dose of 400 mg once daily for 5 consecutive days every 4 weeks.

Azithromycin: an oral dose of 250 mg once daily three times a week (every other day).

Doxycycline: an oral dose of 100 mg once daily.

Placebo will be given as one table once daily.

Study recruitment and enrollment will take place through the Primary Care Research Network (PCRN). Potentially eligible participants aged ≥ 45 will be identified from GP practices up to a 15 mile radius from the RFH. Potential eligible patients will be contacted by letter with an accompanying patient information sheet (PIS) describing the study in detail and inviting the patient to attend a hospital visit and enroll. If patients have not responded to the invitation letter, this will be followed by a reminder letter approximately 2 weeks later. Non responders to the reminder letter will be followed up by a final telephone call. Patients expressing an interest in participation will be offered a screening appointment at the Royal Free Hospital. Patients will be asked to visit the hospital 3 times and will be contacted twice by telephone during the course of the study.

At the Screening Visit (V1), the following will take place:

* The study will be discussed again with the patient during this visit and if he/she agree to participate, they will be asked to sign the consent form.
* A medical history of the patient will be taken. This will include smoking history, antibiotic Hypersensitivity, as well as patient concomitant medication.
* A full physical examination will be performed and height and weight of patients will be recorded.
* A lung function test (spirometry assessment) will be performed.
* A blood sample will be collected in order to perform routine haematology/blood chemistry and liver function.
* A sputum sample will be taken and analysed to determine number of bacteria in the lung and to screen for Tuberculosis.
* A urine pregnancy test will be carried out on females of childbearing potential.
* Patients will be asked to complete two sets of questionnaires; "St. George's respiratory questionnaire" (SGRQ) which includes simple questions about the patients COPD condition and how it affects their life; the second an EQ5D questionnaire which includes simple questions relating to the general quality of their life.
* Patients will be given daily diary cards and asked to record their symptoms.
* An ECG will be performed on all patients.

If patients are eligible for the trial, they will be randomised to one of the following groups:

Moxifloxacin: an oral dose of 400 mg once daily for 5 consecutive days every 4 weeks for a total duration of 13 weeks.

Azithromycin: an oral dose of 250 mg once daily three times a week (every other day) for a total duration of 13 weeks.

Doxycycline: an oral dose of 100 mg once daily, for a total duration of 13 weeks Placebo: an oral daily dose of one capsule, for a total duration of 13 weeks.

This is a single-blind trial. Patients will be blinded to treatment; the investigator will be unblinded. Microbiologists will also be blind to treatment allocation when assessing sputum samples.

Following randomisation of eligible patients, patients will be asked to return to the hospital for a second visit (within 1 week) to collect their medication from the research fellow who will instruct the patient to start taking the medication within 3 days. At this visit, the research team will check if patients are happy filling in their diary cards and will be happy to answer any questions they may have.

In week 5 and week 9 of treatment, each patient will be contacted by telephone to:

* Monitor progress and compliance.
* Remind patients to take medication.
* Encourage patients to contact the GP/investigator if symptoms worsen.
* The occurrence of any adverse effects/serious adverse effects (AE/SAE) or an exacerbation will be checked and recorded.
* Remind patients to fill in their daily diary cards

End of Study Visit (at week 14):

Patients will be asked to return to the hospital and the following assessments will be made:

* The occurrence of AE/SAE or exacerbations will be checked and recorded.
* A spirometry assessment to test their lung function.
* Diary cards will be collected by the investigator.
* SGRQ and EQ5D questionnaires will be completed at this visit by the patient.
* A sputum sample will be taken from the patients to determine bacterial number in their lung.
* Unused study medication and packaging will be collected from the patient.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed COPD diagnosis
* Informed Consent: Patients must give their signed and dated written informed consent to participate
* Gender: Male or female patients
* Age: ≥ 45 years of age at screening
* Produce sputum regularly (produce sputum in at least 3 months of a year)
* Able to complete questionnaires for health status and symptoms and considered able to comply with the dosing regimen.
* Severity of disease: Patients with a measured FEV1<80% of predicted normal values as determined at screening. An average of three spirometry readings will be taken.

Exclusion Criteria:

* Patients with TB, other chronic respiratory disease (e.g. chronic asthma, bronchiectasis, pulmonary fibrosis), patients with hepatic or renal impairment and patients with prolonged QT interval and other cardiac abnormalities.
* Patients with known hypersensitivity to the antibiotics under evaluation.
* Patients on long term antibiotics for other conditions.
* Patients with uncontrolled hypertension.
* Female patients who are pregnant or planning on becoming pregnant during the study, or are breastfeeding.
* Patients with a history of long QT syndrome or whose QTc measured at Visit 1 is prolonged (>450 msec for males and females) as confirmed by the ECG assessor.
* Clinically relevant abnormal laboratory values at the screening assessment that could interfere with the objectives of the trial or safety of the volunteer.
* Patient taking clinically significant contraindicated medication, as per the SmPCs

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-12; Primary Completion 2013-01 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
To measure and compare reduction in the concentration of lower airway bacteria in patients with COPD between three different antibiotic regimes and placebo | Week 14 post treatment

SECONDARY OUTCOMES:
To measure changes in lung function measure, health status and exacerbations. | week 14 post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jadwiga A Wedzicha, Principal Investigator — University College, London
Locations (1):
- Academic Unit of Respiratory Medicine, Royal Free Hospital, London, United Kingdom

REFERENCES:
- [Derived] Brill SE, Law M, El-Emir E, Allinson JP, James P, Maddox V, Donaldson GC, McHugh TD, Cookson WO, Moffatt MF, Nazareth I, Hurst JR, Calverley PM, Sweeting MJ, Wedzicha JA. Effects of different antibiotic classes on airway bacteria in stable COPD using culture and molecular techniques: a randomised controlled trial. Thorax. 2015 Oct;70(10):930-8. doi: 10.1136/thoraxjnl-2015-207194. Epub 2015 Jul 15. PMID 26179246